CLINICAL TRIAL: NCT04053348
Title: Use of Mobile App to Enhance Functional Outcomes and Adherence of Home-based Rehabilitation Program for Elderly With Hip Fracture: A Randomized Controlled Trial
Brief Title: Use of Mobile App to Enhance Geriatric Hip Fracture Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Authority, Hong Kong (Other Government)
Collaborators: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Ken Lau Kin Ming, Physiotherapist I, Hospital Authority, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019.231
Record Dates: First submitted 2019-08-08; First posted 2019-08-12 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Hip Fractures; Rehabilitation
Keywords: Mobile App; Telerehabilitation; Physiotherapy; Hip Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants allocated to the intervention group will receive their home-based rehabilitation program using mobile app installed in the mobile device.
  Interventions: Procedure: Home-based rehabilitation program using mobile app
- Control (Active Comparator): Those assigned to the control group will receive the same home-based rehabilitation program but with information and instructions delivered through the use of paper-based handouts.
  Interventions: Procedure: Home-based rehabilitation program using mobile app

INTERVENTIONS:
Procedure: Home-based rehabilitation program using mobile app — Home-based rehabilitation program
  Other Names: Home-based rehabilitation program using paper-based handouts

SUMMARY:
The steady increase in the incidence of geriatric hip fracture places an increasing burden on health care service in Hong Kong. Post fracture limitations are prominent and restrain many of the elderly from returning to community, rehabilitation is therefore important for reducing their long-term disability.

By integrating the results from pilot application of video guided training and tele-physiotherapy program in different phases of rehabilitation, a Mobile Application (app) is developed aiming to improve hip fracture patients' and their carers' experience throughout the healthcare journey and empower them to manage their own health. A steering group comprised of physiotherapists, informatics and university research expert is formed to co-design the app, compose education content and formulate the promulgation and evaluation strategies. Meetings are also held with all involved clinicians to refine the app before implementation.

This app provides features for hip fracture rehabilitation including "Understanding Hip Fracture", "Hip Fracture Care", "Training" and "Companion". Patients and their carers can obtain hip fracture care related information through the app anywhere, anytime, instead of coming to the clinics in person or reading the information on pamphlets. Physiotherapists can use the app to set training program for discharged patients with "Push Reminder" function and training record can be saved in "Progress Summary", which facilitates them and carers to get a grip on the patients' rehabilitation progress.

Clinical study is therefore planned to be conducted to evaluate the effectiveness of the app from different perspectives, including the users' acceptance and satisfaction, patients' program compliance and functional recovery.

ELIGIBILITY:
Inclusion Criteria:

All participants who completed the inpatient Geriatric Hip Fracture Rehabilitation Program in the Department of Orthopedic Rehabilitation (DOR) of TPH will be recruited by convenience sampling before discharge. To be eligible for enrolment, participants should:

1. have a primary diagnosis of hip fracture,
2. be 60 to 90 years old,
3. be literate enough to read and understand simple questions in Chinese,
4. be discharged home and taken care by caregiver,
5. have at least level III measured by Modified Functional Ambulatory Category (MFAC) upon discharge,
6. have access to a smart phone or tablets (iOS or Android platform)
7. have signed the written informed consent.

Exclusion Criteria:

Participants will be excluded from the study if they:

1. have a bilateral hip fracture or hip fracture is the result of a malignancy,
2. have significant cognitive deficits,
3. have significant cardiopulmonary contraindications or preexisting conditions that precluded participation in an exercise program,
4. have a terminal illness (survival expected to be <1 year),
5. have severe visual deficits or legally blind,
6. have request that their participation be terminated. All eligible participants will be given a detailed explanation and ethics approval will be obtained from the Joint CUHK-NTEC CREC prior to commencing the study.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Lower extremity functional scale | 2 months
  LEFS is a 20-item questionnaire intended to measure patients' functions with a wide range of lower extremity conditions. Each item is rated on a five-point scale (0 - extreme difficulty or unable to perform activity, 4 - no difficulty); total scores range from 0 to 80, and lower scores represent greater difficulty. It has been shown to be highly reliable, correlates with other constructs, and is an independent predictor of patient and physician assessment of change in patients. The minimal clinically important difference (MCID) for the LEFS is 9 points.
Elderly Mobility Scale | 2 months
  The Elderly Mobility scale (EMS) is used to assess an individual's mobility problems through seven functional activities including lying, siting, standing and walking. The possible total score is 20. Patients that get a score under 10 indicate they are dependent in mobility. They require other people to assist their basic activities of daily living (ADL). Patients that get a score between 10 and 13 indicate they are marginal in terms of safe mobility however independent in ADL to a certain extent. Patients that get a score over 14 indicate they are able to perform mobility independently and safely. They are independent in basic ADL. EMS has been demonstrated a good inter-rater reliability and concurrent validity.
Modified Functional Ambulatory Category | 2 months
  The MFAC is a 7-point Likert Scale (1 -7) that is used to classify a patient's walking capacity. Gait is divided into seven categories, ranging from no ability to walk and requires manual assistance to sit or is unable to sit for 1 minute without back or hand support (MFAC 1) to the ability to walk independently on level and non-level surfaces, stairs, and inclines (MFAC 7). The inter-rater reliability of the MFAC (intraclass coefficient [ICC]) was 0.982 (0.971-0.989), with a kappa coefficient of 0.923 and a consistency ratio of 94% for stroke patient and the ICC of the MFAC in patients with hip fractures is 0.96, with a construct validity of r=0.81 on the Elderly Mobility Scale (EMS).
Time Up and Go Test | 2 months
  A test that assesses mobility, balance, walking ability, and fall risk in older adults

SECONDARY OUTCOMES:
Self-reported exercise adherence | 2 months
  Participants will be asked to rate their adherence to their home program using 11-point numerical rating scale (0='never performed my exercises' to 10 = 'always performed my exercises'. This method of capturing adherence is selected because there are few alternative ways of determining adherence that does not involve full-time surveillance.
Exercise logs | 2 months
  Participants will be asked to report their exercise log either by the use of Progress summary function of the app in experimental group or by exercise diaries set out in calendar format prepared in the exercise pamphlet in control group
Modified Caregiver Strain Index | 2 months
  It was designed to detect the physical, psychological, social and financial strain of the informal caregiver. It consisted of 13-items. There were only 3 options (score 2 if the respondent choose "yes", 1 if the respondent choose "yes, sometimes", otherwise score 0 if the respondent choose "no") for the respondent to choose. The CSI score ranged from 0 to 26. Caregivers face a high level of strain if they score high. The modified version of CSI (M-CSI) achieved a high internal reliabilty (α=.90).
System Usability Scale | 2 months
  It is a quick survey to assess the usability of a given product or service. The survey consist ten questions with five possible answers ranging from 'strongly agree' to 'strongly disagree'.
  Scoring SUS
  * For each of the odd numbered questions, subtract 1 from the score.
  * For each of the even numbered questions, subtract their value from 5.
  * Take these new values which you have found, and add up the total score. Then multiply this by 2.5.
  Interpreting Scores The participant's scores for each question are converted to a new number, added together and then multiplied by 2.5 to convert the original scores of 0-40 to 0-100. Though the scores are 0-100, these are not percentages and should be considered only in terms of their percentile ranking.
  Based on research, a SUS score above a 68 would be considered above average and anything below 68 is below average, however the best way to interpret your results involves "normalizing" the scores to produce a percentile ranking.

CONTACTS AND LOCATIONS:
Locations (1):
- Tai Po Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cheng KC, Lau KMK, Cheng ASK, Lau TSK, Lau FOT, Lau MCH, Law SW. Use of mobile app to enhance functional outcomes and adherence of home-based rehabilitation program for elderly with hip fracture: A randomized controlled trial. Hong Kong Physiother J. 2022 Dec;42(2):99-110. doi: 10.1142/S101370252250010X. Epub 2022 Jun 15. PMID 37560168